CLINICAL TRIAL: NCT01226654
Title: Quantitative MR Imaging and Proton Spectroscopy in MS
Brief Title: Quantitative Imaging and Proton Spectroscopy in Multiple Sclerosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 9812; 2R01NS029029-16A1 (NIH)
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Multiple Sclerosis
Keywords: Quantitative Imaging of Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MS Patients (Other): All subjects enrolled in this study will undergo MRI studies. A computerized neuropsychological battery of tests will be administered.
  Interventions: Device: Magnetic Resonance Imaging
- Healthy Patients (Other): Patients enrolled in this study will undergo MRI studies. A computerized neuropsychological battery of tests will be administered.
  Interventions: Device: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Magnetic Resonance Imaging EDSS

SUMMARY:
The primary purpose of this study is to detect changes in the brain that may be associated with multiple sclerosis. Results will be compared to age matched controls. Investigators will assess lesions by measuring T2 and T1 enhanced lesion volumes and magnetization transfer ratio histogram parameters (MTRHP) in patients with relapsing-remitting and secondary-progressive disease. This data will be correlated to total brain parenchymal volume as well as identifying the effect of MS lesions on the gray and white matter, volumetric disability, including Kurtzke Expanded Disability Status Scale (EDSS) and a specific battery of neuropsychological tests. Quantitative analysis of whole brain N-acetylaspartate (WBNAA), a reproducible measure of viable neuron number, using 1H MRS and compare the results to age-matched controls over duration of 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with known MS diagnosis
2. Age 7-110 years
3. Males or females

Exclusion Criteria:

1. Medically unstable
2. Artificial implants in the body
3. Pregnant

Normal Controls

Ages: 7 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 1991-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Assess the MS lesions using Magnetization transfer ratio histogram parameters and compare it to total brain parenchymal volume | 5 years
  1) Lesions will be assessed by measuring T2 and T1 enhanced lesion volumes and magnetization transfer ratio histogram parameters (MTRHP) in patients with relapsing-remitting and secondary-progressive disease. This data will be correlated to total brain parenchymal volume as well as identifying the effect of MS lesions on the gray and white matter, volumetric disability, including Kurtzke Expanded Disability Status Scale (EDSS) and a specific battery of neuropsychological tests

SECONDARY OUTCOMES:
Quantitative analysis of whole brain N-acetylaspartate (WBNAA) | 5 years
  Quantitative analysis of whole brain N-acetylaspartate (WBNAA), a reproducible measure of viable neuron number, using 1H MRS and compare the results to age-matched controls over duration of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yulin Ge, M.D., Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

REFERENCES:
- [Result] Ge Y, Zohrabian VM, Osa EO, Xu J, Jaggi H, Herbert J, Haacke EM, Grossman RI. Diminished visibility of cerebral venous vasculature in multiple sclerosis by susceptibility-weighted imaging at 3.0 Tesla. J Magn Reson Imaging. 2009 May;29(5):1190-4. doi: 10.1002/jmri.21758. PMID 19388109